CLINICAL TRIAL: NCT06025838
Title: Positive Feedback vs. No-Feedback Games for Behavioral Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bard College (Other)
Responsible Party: Principal Investigator, Justin Dainer-Best, Associate Professor of Psychology, Bard College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FeedbackGames
Record Dates: First submitted 2023-08-30; First posted 2023-09-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder; Low Mood
MeSH Terms: conditions — Depressive Disorder, Major; Consciousness Disorders | interventions — Feedback, Physiological

STUDY DESIGN:
Intervention Model Description: Participants are either assigned to a control (no intervention) condition or to one where they receive positive feedback and are encouraged to specific, positive behavior.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention occurs entirely online. All assessment occurs via survey software. Participants do not interact with other participants and are not fully informed of the nature of the intervention and thus do not know if they are in an active condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- positive feedback (Experimental): Participants receive positive feedback and reward for their decisions taken during a small game similar to a normal person's life. For example, they are encouraged to exercise, make food, and interact with friends.
  Interventions: Behavioral: positive feedback
- no feedback (No Intervention): Participants receive no feedback. While they may undertake the same decisions during a small game similar to a normal person's life, they receive no encouragement and are not given reward or positive feedback.

INTERVENTIONS:
Behavioral: positive feedback — The positive feedback game uses techniques relating to established therapies like Behavioral Activation and Acceptance and Commitment Therapy's valued living to encourage positive action in game and outside of the game.
  Arms: positive feedback

SUMMARY:
We aim to investigate here whether we can develop a reinforcement learning game which provides game-based feedback to encourage positive actions (behaviors) both inside and outside of the game. Does providing positive reward when participants make decisions which are associated with value-based actions (like those in BA) result in different game decisions? We propose that it will increase positive actions in the game. And, secondly, how does it affect short-term behavior (in one week)? We propose that it will increase pro-health activities and may reduce depressive symptoms.

DETAILED DESCRIPTION:
We know that behavior influences mood -- our best interventions to improve mood rely upon the relationship between these. Treatments like this are thought to work in part by helping individuals to increase value-derived behaviors; participants are given guidance which results in an increase of positive behaviors and a decrease of coping behaviors that don't help -- that is, their health-seeking behavior is reinforced while behaviors that diminish health are reduced. In past work, we showed that a text-based game could be used to explore what sort of decisions people would make in certain environments. That game showed associations between in-game behaviors and real-life depressive symptoms and actions. Such work focuses on low-level symptoms of depression -- increasingly common, especially after the onset of the covid-19 pandemic. We aim to investigate here whether we can develop a reinforcement learning game which provides game-based feedback to encourage positive actions (behaviors) both inside and outside of the game.

Thus, the experiment described below and proposed in this application would test the role of positive rewards (positive-feedback) in a dichotomous-choice game, compared to neutral (no-feedback).

ELIGIBILITY:
Inclusion Criteria:

* 18-34 years old
* Fluent in English
* Based in the United States

Exclusion Criteria:

* None

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-8 item) | baseline (T0) - before intervention
  8 items rated in a self-report questionnaire. Scores range from 0 to 24 with higher scores indicating more depression symptoms.
Depressive symptoms (Patient Health Questionnaire-8 item) | one week following intervention (T1)
  8 items rated in a self-report questionnaire. Scores range from 0 to 24 with higher scores indicating more depression symptoms.
Day Reconstruction Method (DRM) | baseline (T0) - before intervention
  The DRM measures how people spend their time and asks them how they felt while doing the activities they report. Ratings on a Likert scale indicate valence (how pleasant/unpleasant the activities were) and range from 0 (not at all) to 6 (very much), with higher pleasantness being better (and lower unpleasantness being better).
Day Reconstruction Method (DRM) | one week following intervention (T1)
  The DRM measures how people spend their time and asks them how they felt while doing the activities they report. Ratings on a Likert scale indicate valence (how pleasant/unpleasant the activities were) and range from 0 (not at all) to 6 (very much), with higher pleasantness being better (and lower unpleasantness being better).
Behavior in study-specific game | baseline (T0)
  For both conditions, behavior and choices made during the game will be used as data for analyses. Game choices allow participants to decide what next activities they will "do" in the game. Analyses incorporate decision probabilities (which of 2 choices are selected) and compare them between conditions. The game is completed at baseline following assessment.
Motivation to change | baseline (T0) - after intervention
  A 7-point item, "It is important to me to do more positive activities in my life". Scores range from 0 [not at all] to 6 [very much]. Higher scores indicate more motivation to change.

SECONDARY OUTCOMES:
Mood and Anxiety Symptoms Questionnaire (MASQ) | baseline (T0) - before intervention
  The MASQ measures mood and anxiety symptoms on three subscales: Anhedonic Depression, Anxious Arousal, and General Distress. Scores on each subscale range from 10 (low symptoms) to 50 (high symptoms). Higher scores indicate more depression, anxiety, and distress.
Mood Ratings | baseline (T0) - before intervention
  Mood will be rated on positive and negative scales: "On the whole, how sad were you today?" (Rated from 0 [not at all] to 6 [extremely]); "On the whole, how happy were you today?" (Rated from 0 [not at all] to 6 [extremely]). Higher scores indicate more sadness or happiness.
Mood Ratings | one week following intervention (T1)
  Mood will be rated on positive and negative scales: "On the whole, how sad were you today?" (Rated from 0 [not at all] to 6 [extremely]); "On the whole, how happy were you today?" (Rated from 0 [not at all] to 6 [extremely]). Higher scores indicate more sadness or happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Dainer-Best, Ph.D., Principal Investigator — Bard College
Locations (1):
- Online research conducted through Bard College, Annandale-on-Hudson, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on the Open Science Framework, https://osf.io
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available on or before a manuscript is submitted for publication and will be shared indefinitely.
Access Criteria: Open access. Anyone will be able to access de-identified data and code.
URL: https://doi.org/10.17605/osf.io/y893q